CLINICAL TRIAL: NCT06307158
Title: Influence of Intraoperative Blood Salvage and Autotransfusion on Tumor Recurrence After Deceased Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2024-ZJU-OBS1
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intraoperative blood salvage and autotransfusion (IBSA) group: The study included patients who underwent adult-to-adult DDLT for HCC in China between January 2015 and December 2020. Exclusion criteria included: patients under 18 years of age, presence of extrahepatic metastasis, combined kidney transplantation, reduced-size or split liver transplantation, re-transplantation, and missing data on analyzed variables. The remaining recipients were 349 in IBSA group who received salvaged blood autotransfusion during the LT.
- non-intraoperative blood salvage and autotransfusion (non-IBSA) group: The study included patients who underwent adult-to-adult DDLT for HCC in China between January 2015 and December 2020. Exclusion criteria was as mentioned ahead. Recipients who did not receive salvaged blood autotransfusion during the LT were enrolled in non-IBSA group.

SUMMARY:
The practice of intraoperative blood salvage and autotransfusion (IBSA) during deceased donor liver transplantation (DDLT) for hepatocellular carcinoma (HCC) can potentially reduce the need for allogeneic blood transfusion. However, implementing IBSA remains debatable due to concerns about its possible detrimental effects on oncologic recurrence. Hence, a nationwide multi-center study was conducted to investigate further the association between IBSA and post-transplant HCC recurrence, including a stratified subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult-to-adult deceased donor liver transplantation for hepatocellular carcinoma

Exclusion Criteria:

* patients under 18 years of age
* presence of extrahepatic metastasis
* combined kidney transplantation
* reduced-size or split liver transplantation
* re-transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective review was conducted on the prospectively maintained liver transplantation database of the CLTR. The initial data collection included patients who underwent adult-to-adult DDLT for HCC in China between January 2015 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative recurrence of liver cancer | 2015.1.1-2020.12.31
  The overall incidence of HCC recurrence (intrahepatic or extrahepatic) after LT.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang M, Wei X, Shu W, Zhai X, Zhou Z, Cai J, Yang J, Jin B, Zheng S, Xu X. Influence of intraoperative blood salvage and autotransfusion on tumor recurrence after deceased donor liver transplantation: a large nationwide cohort study. Int J Surg. 2024 Sep 1;110(9):5652-5661. doi: 10.1097/JS9.0000000000001683. PMID 38847771